CLINICAL TRIAL: NCT06846398
Title: A Phase 2, Open-label, Multicenter Study to Assess the Efficacy and Safety of BW-20805 in Adult Subjects With Hereditary Angioedema
Brief Title: A Phase 2 in Adult Subjects With Hereditary Angioedema
Acronym: HAE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Argo Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BW-20805-2001
Record Dates: First submitted 2025-02-13; First posted 2025-02-26 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Hereditary Angioedema (HAE)
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Experimental): BW-20805 600 mg Q24W*2
  Interventions: Drug: BW-20805
- Cohort 2 (Experimental): BW-20805 300 mg Q24W*2
  Interventions: Drug: BW-20805
- Cohort 3 (Experimental): BW-20805 300 mg Q12W*2
  Interventions: Drug: BW-20805

INTERVENTIONS:
Drug: BW-20805 — SC administrations of BW-20805 600 mg on Day1 to Day673
  Arms: Cohort 1
Drug: BW-20805 — SC administrations of BW-20805 300 mg every 24 weeks on Day1 to Day169;Day337 to Day673
  Arms: Cohort 2
Drug: BW-20805 — SC administrations of BW-20805 300 mg every 12 weeks on Day 1 to Day 589
  Arms: Cohort 3

SUMMARY:
A Phase 2 in Adult Subjects with Hereditary Angioedema

DETAILED DESCRIPTION:
A Phase 2, Open-label, Multicenter Study to Assess the Efficacy and Safety of BW-20805 in Adult Subjects with Hereditary Angioedema

ELIGIBILITY:
Inclusion Criteria:

* Must have given written informed consent and be able to comply with all study requirements.
* Males or females 18 to 70 years of age at the time of informed consent.
* Documented diagnosis of HAE-1/HAE-2.
* At least 2 HAE attacks within the 8-week run-in period, as confirmed by an investigator based on the protocol-specified definition
* Access to and ability to use ≥ 1 acute medication(s)
* Female subjects must be non-pregnant;non-lactating, and either surgically sterile
* Male subjects with WOCBP partners, dual contraception is required if no surgically sterile

Exclusion Criteria:

* Any clinically significant medical or psychiatric condition or medical history that, in the opinion of the Investigator, makes the subject unsuitable for participation in the study
* Any concomitant diagnosis of another form of chronic angioedema, such as acquired angioedema, HAE with normal C1-INH, idiopathic angioedema, or recurrent angioedema associated with urticaria
* History or presence of carcinoma within 5 years prior to screening, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated.
* Have undergone major surgery within 3 months prior to screening.
* History of clinically significant arterial or venous thrombosis, or current clinically significant prothrombotic or bleeding risk
* History of allergic reaction to an oligonucleotide or N-acetylgalactosamine
* Prior treatment with any oligonucleotides within 6 months if single dose or 12 months if multiple doses prior to screening.
* Exposure to another investigational drug or biological agent within 30 days or within at least 5 half-lives prior to screening.
* With ANY of the abnormalities in clinical laboratory tests at screening and run-in period
* Clinically significant findings on 12-lead electrocardiogram that would place the patient at risk or interfere with participation in the study at screening.
* Positive for Human immunodeficiency virus (HIV), HBsAg, Hepatitis C or syphilis infection
* Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to dosing.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
To determine the prophylactic effect of in HAE attack rate. | from baseline to Day169
  Change in time-normalized monthly (per 4 weeks) HAE attack rate from baseline to Day169

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of multiple doses of BW-20805. | up to 96 weeks
  Incidence and severity of SAEs and AEs up to 96 weeks ( the main study period, extension study period and whole study)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Magerl, Doctor, Principal Investigator — Charite-Universitaetsmedizin Berlin - Klinik fuer Dermatologie Venerologie und Allergologie
Locations (18):
- United States (5):
  - Institute for Asthma and Allergy - Wheaton, Silver Spring, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University Medicine Center, Durham, North Carolina
  - Penn State Milton S. Hershey MC - Penn State, Hershey, Pennsylvania
  - Inova Clinical Trials and Research Center, Falls Church, Virginia
- China (6):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - West China Hospital, Sichuan University, Chengdu, Sichaun
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
- Germany (2):
  - Universitätsmedizin der Johannes Gutenberg, Mainz, Rhineland-Palatinate
  - Charité - Universitätsmedizin Berlin, Berlin, State of Berlin
- Italy (3):
  - Azienda Ospedaliero Universitaria Policlinico G. Rodolico San Marco - Ospedale San Marco, Catania, Catania
  - Azienda Ospedaliero-Universitaria Careggi, Florence, Florence
  - Azienda Ospedale - Universita di Padova, Padua, PD
- SP ZOZ Szpital Uniwersytecki w Krakowie, Krakow, Lesser Poland Voivodeship, Poland
- Hospital Universitario Virgen del Rocío, Seville, Sevilla, Spain

IPD SHARING:
Plan to Share IPD: No